CLINICAL TRIAL: NCT01754623
Title: Validation of a Radiation Response Signature in Borderline Resectable Pancreatic Cancer Patients Treated With Induction Chemotherapy Followed by Stereotactic Body Radiation Therapy (SBRT)
Brief Title: GTX-RT in Borderline Resectable Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of pre-treatment tissue to make the study plan feasible.
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16932
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-06

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas; Pancreatic; Neoplasms; Stereotactic; Radiosurgery; Borderline; Resectable; Gastrointestinal; Gemcitabine; Capecitabine; Fluorouracil; Docetaxel; SBRT; GTX Chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Capecitabine; Gemcitabine; Docetaxel; Radiosurgery; Surgical Procedures, Operative; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy Followed by Radiation Treatment (Experimental): Gemcitabine, Taxotere, Xeloda (GTX): 21 day cycle x 3 Gemcitabine 750mg/m^2 on days 4 and 11 Taxotere® (docetaxel) 30 mg/m^2 on days 4 and 11 Xeloda® (capecitabine) 750 mg/m^2 on days 1-14 Radiation: stereotactic body radiation therapy stereotactic body radiation therapy (SBRT).
  After radiation, participants will be re-evaluated for surgery.
  Interventions: Drug: Capecitabine; Drug: Gemcitabine; Drug: Docetaxel; Radiation: Stereotactic body radiation therapy (SBRT); Other: Restaging review after radiation; Procedure: Surgery; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Capecitabine — Treatment will begin with the first round of chemotherapy. Each round of chemotherapy will take 21 days. Each round or cycle will start with participants taking capecitabine pills. Participants will take tablets of capecitabine (Xeloda®) twice per day for 14 days followed by 7 days without capecitabine.
  Other Names: Xeloda®
Drug: Gemcitabine — On the fourth day of the cycle, participants will be treated with gemcitabine and docetaxel. First, this will consist of placing gemcitabine (Gemzar®) in a bag of fluid and giving it by vein over 30 minutes.
  Other Names: Gemzar®
Drug: Docetaxel — On the fourth day of the cycle, participants will be treated with gemcitabine and docetaxel. After the gemcitabine, participants will receive docetaxel (Taxotere®) in a bag of fluid over 1 hour.
  Other Names: Taxotere®
Radiation: Stereotactic body radiation therapy (SBRT) — 30/40 Gy to pancreatic tumor/area of borderline resectability
  Other Names: SBRT
Other: Restaging review after radiation — After radiation, participants will be re-evaluated for surgery. Patients who have Complete Response (CR), Partial Response (PR) or stable disease (SD) will proceed with surgical exploration and resection provided they are suitable fit for surgery in the judgment of the surgical oncologist. Patients who have local progression on imaging scan will be offered conventional 5-Fluorouracil based intensity-modulated radiation therapy (IMRT). If no surgery: then chemotherapy. If surgery: chemotherapy will be given based on response.
Procedure: Surgery — Non-metastatic patients who are deemed resectable after neoadjuvant therapy will be taken to surgery. After surgery, chemotherapy will be given based on response.
Drug: 5-Fluorouracil — Patients who have local progression on imaging scan will be offered conventional 5-Fluorouracil based intensity-modulated radiation therapy (IMRT).

SUMMARY:
The purpose of this study is to find out if a program of intensive chemotherapy with gemcitabine, docetaxel and capecitabine followed by an advanced form of focused radiation aimed at participant's tumor followed by more chemotherapy can increase the chances that the participant's pancreatic tumor can be removed completely.

DETAILED DESCRIPTION:
Investigators plan to conduct a prospective pilot phase II trial of GTX-SBRT as neoadjuvant treatment of borderline resectable pancreatic cancer. After informed consent, pretreatment pancreatic tumor tissues will be collected and immediately frozen at the time of staging endoscopic ultrasound (EUS). Ribonucleic acid (RNA) will be extracted from tumor specimens and run on microarray analysis to determine radiosensitivity index score. Borderline resectable (BR) patients will be treated with 3 cycles of GTX chemotherapy followed by SBRT. They will be restaged and evaluated for resectability 3 to 4 weeks later. Non-metastatic patients who are deemed resectable after neoadjuvant therapy will be taken to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed pancreatic adenocarcinoma that is borderline resectable disease. Borderline resectable lesions are defined as:

  * circumferential tumor abutment with the superior mesenteric vein (SMV) or portal vein (PV) or SMV/PV confluence over </= 180°
  * circumferential tumor abutment with the superior mesenteric artery (SMA) over </= 180°
  * Short segment encasement (360°) of the PV or SMV that is amenable to partial vein resection and reconstruction
  * encasement of the gastroduodenal artery up to the origin of the hepatic artery
* Patients must have measurable disease
* No previous chemotherapy or radiation to the pancreas
* Eastern Cooperative Oncology Group (ECOG) performance status </= 2 (Karnofsky >/= 60%)
* Patients must have normal organ and marrow function as defined below:

  * leukocytes >/= 3,000/μL
  * absolute neutrophil count >/= 1,000/ μL
  * platelets >/= 100,000/ μL
  * creatinine within normal institutional limits (ULN)
  * total bilirubin will allow for 2x the upper limit of the institution. Patients may have biliary stents or drains to lower total bilirubin to this range.
* Has a negative serum or urine pregnancy test within 7 days prior to initiation of therapy (female patients of childbearing potential). Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Patients will agree to continue contraception for 30 days from the date of the last study drug administration.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with metastatic disease are ineligible.
* Patients who have had prior chemotherapy for pancreatic adenocarcinoma
* Patients who have received prior radiation to an abdominal site are not eligible.
* Patients with peripheral neuropathy >/= grade 2
* Patients with a history of severe hypersensitivity reaction to Taxotere (docetaxel), other drugs formulated with polysorbate 80, gemcitabine, or capecitabine
* Patients may not be receiving any other investigational agents.
* ECOG Performance Status 3-4
* Pregnant or breast-feeding women are excluded from this study because gemcitabine,capecitabine, and docetaxel are Class D agents with the potential for teratogenic or abortifacient effects.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not have any comorbid inflammatory conditions of the bowel such as Crohn's Disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Shridhar, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Strom T, Hoffe SE, Fulp W, Frakes J, Coppola D, Springett GM, Malafa MP, Harris CL, Eschrich SA, Torres-Roca JF, Shridhar R. Radiosensitivity index predicts for survival with adjuvant radiation in resectable pancreatic cancer. Radiother Oncol. 2015 Oct;117(1):159-64. doi: 10.1016/j.radonc.2015.07.018. Epub 2015 Jul 30. PMID 26235848

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center from March 2013 through December 2013.
Period: Overall Study
Arm/Group | Chemotherapy Followed by Radiation Treatment
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Chemotherapy Followed by Radiation Treatment
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Margin-negative (R0) Resection Rate
Description: R0 rate for all participants with resection. Margin negative surgery (R0 resection) is an absolute part of the curative treatment of pancreatic cancer.The primary endpoint is correlation of a radio sensitivity index score derived from the microarray analysis and pathologic response on surgical specimens. Tumor regression Rating: R0 (Complete Response). R0 resections are scored as those resections in which the common bile duct margin, pancreatic resection margin, retroperitoneal margin are negative for tumor involvement.
Time Frame: Up to 3 years
Population: All participants with resection
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy Followed by Radiation Treatment
Number analyzed (Participants) | 3
percentage of participants | 67

2. Secondary Outcome: Progression-Free Survival (PFS) at Three Years
Description: PFS is defined as the duration of time from enrollment to time of death or progression of disease, whichever occurs first. Progressive Disease (PD): At least a 20% increase in the longest diameter (LD) of the target lesion or appearance of new lesions at metastatic sites.
Time Frame: 3 years
Population: Evaluable participants at 3 years.
Arm/Group | Chemotherapy Followed by Radiation Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival (OS) Rate
Description: OS at time of analysis, calculated from date of enrollment to date of death from any cause.
Time Frame: 12 months
Population: All participants per group
Measure: Number; unit: percentage of participants
Groups:
- All Participants -Chemotherapy Followed by Radiation Treatment; Resection Group -Chemotherapy Followed by Radiation Treatment: Gemcitabine, Taxotere, Xeloda (GTX): 21 day cycle x 3 Gemcitabine 750mg/m^2 on days 4 and 11 Taxotere® (docetaxel) 30 mg/m^2 on days 4 and 11 Xeloda® (capecitabine) 750 mg/m^2 on days 1-14 Radiation: stereotactic body radiation therapy stereotactic body radiation therapy (SBRT).
  After radiation, participants will be re-evaluated for surgery.
Arm/Group | All Participants -Chemotherapy Followed by Radiation Treatment | Resection Group -Chemotherapy Followed by Radiation Treatment
Number analyzed (Participants) | 9 | 3
percentage of participants | 33 | 100

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Arm/Group | Chemotherapy Followed by Radiation Treatment
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy Followed by Radiation Treatment (N=9)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disorders - Other, Liver abscess (Hepatobiliary disorders) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy Followed by Radiation Treatment (N=9)
Diarhea (Gastrointestinal disorders) | 6 (9)
Constipation (Gastrointestinal disorders) | 5 (6)
Abdmonimal pain (Gastrointestinal disorders) | 2 (4)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 9 (13)
Fever (General disorders) | 2 (2)
Flu like symptoms (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (2)
Irritability (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (8)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3)
Palmar-plantar erthrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Tegaderm skin reaction from IV (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 6 (14)
Neutrophil count decreased (Investigations) | 3 (5)
Platelet count decreased (Investigations) | 3 (8)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 2 (5)
Blood bilirubin increased (Investigations) | 1 (2)
CD4 lymphocytes decreased (Investigations) | 1 (4)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Pancreatic enzymes (Investigations) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Depressioin (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Hallucinations (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 3 (4)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study only accrued 9 (of planned 35) participants. It was not possible to collect adequate pre-treatment tissue for radiosensitivity index (RSI) analysis, pre-treatment. The study was terminated before planned completion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No